CLINICAL TRIAL: NCT03002857
Title: Comparison of I-gel LMA, Classical LMA With a New Supraglottic Airway the Baska Mask®in Urological Surgery Regarding Their Efficacy and Safety
Brief Title: Comparison of I-gel LMA, Classical LMA With a New Supraglottic Airway the Baska Mask® in Urological Surgery
Acronym: BCIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Collaborators: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Ülkü Sabuncu, M.D., Adiyaman University Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: LMA-Urological surgery
Record Dates: First submitted 2016-12-17; First posted 2016-12-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Airway Management
Keywords: Laryngeal Mask Airway; Urologic Surgical Procedure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Classical LMA (Experimental): Classical LMA insertion: LMA-C insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and end-tidal carbon dioxide pressure waveform.
  Interventions: Device: LMA-C
- I-gel (Experimental): I-gel LMA insertion: The I-gel LMA insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and end-tidal carbon dioxide pressure waveform.
  Interventions: Device: I-gel
- The Baska Mask® (Experimental): The Baska Mask® insertion: The Baska Mask® insertion was done in supine position and with a standard gel pillow with the patient's head on following anesthesia induction. The insertion was verified with the manual ventilation of the patient and end-tidal carbon dioxide pressure waveform.
  Interventions: Device: Baska Mask

INTERVENTIONS:
Device: LMA-C — LMA-C will be placed into the patients airway following anesthesia induction. The placement will be done as suggested in supine position with a standard gel pillow under patients head.
  Arms: Classical LMA
Device: Baska Mask — Baska Mask will be placed into the patients airway following anesthesia induction. The placement will be done as suggested in supine position with a standard gel pillow under patients head.
  Arms: The Baska Mask®
Device: I-gel — I-gel LMA placement will be done as suggested in supine position with a standard gel pillow under patients head.
  Arms: I-gel

SUMMARY:
The most used airway management strategies are different types of supraglottic airway devices (SAD) for transurethral resection of bladder and ureteroscopy in urological surgery . Classical laryngeal mask airway (LMA-C) and I-Gel SADs are being used already. The aim of this study was to evaluate and compare the performance of a new type of SAD the Baska Mask® with I-gel and LMA-C regarding their insertion times, durations, perioperative complications and effects on hemodynamic parameters, peak airway pressures (Paw) and airway plato pressures in urological surgery as well.

DETAILED DESCRIPTION:
The most used airway management strategies are different types of supraglottic airway devices (SAD) for transurethral resection of bladder and ureteroscopy in urological surgery . Classical laryngeal mask airway (LMA-C) and I-Gel SADs are being used already. The aim of this study was to evaluate and compare the performance of a new type of SAD the Baska Mask® with I-gel and LMA-C regarding their insertion times, durations, perioperative complications and effects on hemodynamic parameters, peak airway pressures (Paw) and airway plato pressures in urological surgery as well.

The main suggestion about the Baska Mask® is that it's the most appropriate airway device with high Paws. In high Paws, higher air leaks may occur from the sides of cuff and this causes hypoventilation. So the main aim of this study is to evaltuate three devices in terms of insertion and ventilation times, the "first attempt" success rates, the additional maneuvering requirements and complications developed after intervention.

The secondary objective of the study was to evaluate all three SADs in terms of airway pressures producing sufficient tidal volume and hemodynamical parameters.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) 1-2-3 physical status scheduled for elective surgical procedure for transurethral resection of bladder and ureteroscopy.

Exclusion Criteria:

* Under the age of 18, history of hiatus hernia, gastroesophageal reflux, body mass index (BMI) > 30 kg m-2, ASA physical status 4 or over and patients who met the difficult intubation criteria.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Insertion times | Perioperative
  It was evaluated that how many secs does it take to insert properly.
Ventilation times | Perioperative
  It was evaluated that how many secs does it take to ventilate the patient.
First attemp success rates | Perioperative
  In how many patients it was inserted at first attempt
The additional maneuvering | Perioperative
  ıt was evaluated how many maneuvers needed to insert the device.
Airway related complications | Perioperative
  Complications like Bloodstain of the mask, Dysphagia, Tongue injury, Lips injury, Teeth injury, Palate injury, Sore throat, Hoarseness, Desaturation , Laryngospasm, Regurgitation/aspiration were evaluated.

SECONDARY OUTCOMES:
Airway PAP and Plateau pressures | Perioperative
  Both pressures were evaluated following device insertion and then in every 10 mins.
Haemodynamic parameters, heart rate bpm, systolic and diastolic arterial pressures mmHg | Perioperative
  Preoperative and following device insertion all haemodynamic parameters were evaluated in every 10 mins.

CONTACTS AND LOCATIONS:
Overall Officials: Asli Demir, Study Director — Yuksek Ihtisas Research and Educational Hospital

IPD SHARING:
Plan to Share IPD: No